CLINICAL TRIAL: NCT00490815
Title: An Open Label Pharmacokinetic and Efficacy Study of 0.5 μg/Day and 0.2 μg/Day Fluocinolone Acetonide Intravitreal Inserts in Subjects With Diabetic Macular Edema
Brief Title: Pharmacokinetic and Efficacy Study of Fluocinolone Acetonide Inserts in Patients With Diabetic Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alimera Sciences (Industry)
Responsible Party: Sponsor
Organization: ANI Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-01-06-002
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Results first posted 2014-02-13 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Fluocinolone Acetonide

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Fluocinolone Acetonide
- 2 (Experimental)
  Interventions: Drug: Fluocinolone Acetonide

INTERVENTIONS:
Drug: Fluocinolone Acetonide — 0.5 mg fluocinolone acetonide intravitreal insert
  Arms: 1
Drug: Fluocinolone Acetonide — 0.2 mg fluocinolone acetonide intravitreal insert
  Arms: 2

SUMMARY:
This study will evaluate the pharmacokinetics, safety and efficacy of an intravitreal insert of fluocinolone acetonide for the treatment of diabetic macular edema

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years with diabetic macular edema
* Diagnosis of diabetes mellitus types 1 or 2
* Best corrected visual acuity of ≥ 19 letters
* Retinal thickness > 250 microns by OCT
* Investigator is comfortable deferring macular laser treatment for 6 weeks

Exclusion Criteria:

* Glaucoma, ocular hypertension, IOP >21 mmHg or concurrent therapy at screening with IOP lowering agents
* Retinal or choroidal neovascularization due to ocular conditions other than diabetic retinopathy
* Prior intravitreal, subtenon, or periocular steroid therapy within the last 3 months
* Prior intravitreal or subtenon anti-VEGF therapy within the last 2 months
* Any ocular surgery within the last 3 months
* Retinal laser treatment within the last 3 months
* History of uncontrolled IOP elevation with steroid use that did not respond to topical therapy
* Any lens opacity which impairs visualization of the posterior pole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-08; Primary Completion 2009-09 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- John Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluocinolone Acetonide: 0.2 ug/Day Implant: Dose 0.2 ug/day Medidur Implant administered in one eye
- Fluocinolone Acetonide: 0.5 ug/Day Implant: Dose 0.5 ug/day Medidur Implant administered in one eye
Period: Overall Study
Arm/Group | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant
Started | 20 | 17
Completed | 12 | 8
Not Completed | 8 | 9
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Death | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Fluocinolone Acetonide: 0.2 ug/Day Implant: Dose 0.2 ug/day Medidur Implant
- Fluocinolone Acetonide: 0.5 ug/Day Implant: Dose 0.5 ug/day Medidur Implant
- Total: Total of all reporting groups
Arm/Group | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (9.4) | 67.4 (10.3) | 66.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 10 | 11 | 21
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Levels of Fluocinolone Acetonide in Plasma and Aqueous Humor
Description: This was a combined assessment of the levels of fluocinolone acetonide in the plasma and aqueous humor. The average values of the data collected is entered in Outcome Data.
Time Frame: over 36 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant
Number analyzed (Participants) | 12 | 8
pg/ml | 1.4905 (1.87058) | 0.7140 (0.78096)

2. Secondary Outcome: Retinal Thickness
Time Frame: over 36 months
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant
Number analyzed (Participants) | 20 | 17
µg | 343.8 (142.92) | 324.2 (136.86)

ADVERSE EVENTS:
Arm/Group | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant
Serious Adverse Events (participants affected / at risk) | 19/20 | 12/17
Other Adverse Events (participants affected / at risk) | 20/20 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluocinolone Acetonide: 0.2 ug/Day Implant (N=20) | Fluocinolone Acetonide: 0.5 ug/Day Implant (N=17)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 2 (2) — #Study eye
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 13 (13) | 5 (5) — #Study eye
Cataract operation (Surgical and medical procedures) | 5 (5) | 4 (4) — #Fellow eye
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Colectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Glaucoma surgery (Surgical and medical procedures) | 0 (0) | 2 (2) — #Study eye
Retinal operation (Surgical and medical procedures) | 1 (1) | 0 (0) — #Study eye
Retinal operation (Surgical and medical procedures) | 1 (1) | 0 (0) — #Fellow eye
Trabeculectomy (Surgical and medical procedures) | 1 (1) | 2 (2) — #Study eye
Vitrectomy (Surgical and medical procedures) | 1 (1) | 0 (0) — #Study eye
Vitrectomy (Surgical and medical procedures) | 1 (1) | 0 (0) — #Fellow eye
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluocinolone Acetonide: 0.2 ug/Day Implant (N=20) | Fluocinolone Acetonide: 0.5 ug/Day Implant (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Asthenopia (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Asthenopia (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Cataract (Eye disorders) | 11 (11) | 4 (4) — #Study eye
Cataract (Eye disorders) | 6 (6) | 4 (4) — #Fellow eye
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Cataract subcapsular (Eye disorders) | 1 (1) | 3 (4) — #Study eye
Conjunctival haemorrhage (Eye disorders) | 7 (8) | 7 (9) — #Study eye
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Corneal oedema (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Diabetic retinal oedema (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Diplopia (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Diplopia (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Dry eye (Eye disorders) | 1 (1) | 2 (2) — #Study eye
Dry eye (Eye disorders) | 1 (1) | 2 (2) — #Fellow eye
Eye irritation (Eye disorders) | 1 (3) | 2 (2) — #Study eye
Eye irritation (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Eye pain (Eye disorders) | 4 (4) | 2 (5) — #Study eye
Eye pain (Eye disorders) | 3 (3) | 0 (0) — #Fellow eye
Eye pruritus (Eye disorders) | 2 (3) | 1 (1) — #Study eye
Eye pruritus (Eye disorders) | 1 (2) | 0 (0) — #Fellow eye
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Foreign body sensation in eyes (Eye disorders) | 2 (2) | 1 (1) — #Study eye
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Glaucoma (Eye disorders) | 1 (1) | 1 (2) — #Study eye
Iris atrophy (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Iris neovascularisation (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Lacrimation increased (Eye disorders) | 1 (1) | 1 (1) — #Study eye
Lacrimation increased (Eye disorders) | 1 (1) | 3 (3) — #Fellow eye
Macular hole (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Macular ischaemia (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Maculopathy (Eye disorders) | 4 (5) | 0 (0) — #Study eye
Maculopathy (Eye disorders) | 2 (2) | 1 (1) — #Fellow eye
Myodesopsia (Eye disorders) | 7 (10) | 6 (11) — #Study eye
Myodesopsia (Eye disorders) | 1 (1) | 1 (1) — #Fellow eye
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Ocular hyperaemia (Eye disorders) | 1 (1) | 2 (2) — #Study eye
Optic atrophy (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Optic atrophy (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Photophobia (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Photopsia (Eye disorders) | 1 (1) | 1 (1) — #Study eye
Posterior capsule opacification (Eye disorders) | 2 (3) | 1 (1) — #Study eye
Posterior capsule opacification (Eye disorders) | 0 (0) | 1 (1) — #Fellow eye
Retinal aneurysm (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Retinal vascular occlusion (Eye disorders) | 1 (1) | 0 (0) — #Study eye
Vision blurred (Eye disorders) | 1 (1) | 1 (1) — #Study eye
Vision blurred (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Visual impairment (Eye disorders) | 0 (0) | 2 (2) — #Study eye
Vitreous detachment (Eye disorders) | 2 (2) | 1 (1) — #Study eye
Vitreous haemorrhage (Eye disorders) | 3 (3) | 1 (5) — #Fellow eye
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Blister infected (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (2) | 0 (0) — #Study eye
Hordeolum (Infections and infestations) | 1 (2) | 0 (0) — #Fellow eye
Infected bites (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cataract operation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — #Study eye
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — #Study eye
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 2 (3)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — #Study eye
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 4 (5) | 7 (12) — #Study eye
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) — #Fellow eye
Optic nerve cup/disc ratio increased (Investigations) | 1 (1) | 0 (0) — #Study eye
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (3) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Visual field defect (Nervous system disorders) | 1 (1) | 0 (0) — #Study eye
Anticipatory anxiety (Psychiatric disorders) | 0 (0) | 1 (3)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergic respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — #Study eye
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days